CLINICAL TRIAL: NCT05973045
Title: Investigation of the Effect of Distention Medium Temperature on Image Quality, Hyponatremia Risk and Post-operative Pain in Operative Hysteroscopy
Brief Title: Investigation of the Effect of Distention Medium Temperature on Image Quality, Hyponatremia Risk, and Post-operative Pain in Operative Hysteroscopy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Sabahattin Anıl Arı, Asst. Prof., Izmir Bakircay University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 617
Record Dates: First submitted 2023-07-25; First posted 2023-08-02 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Post-operative Pain
Keywords: hysteroscopy
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Prospective Randomized Controlled Clinical Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 24 Centigrade Degree (Active Comparator): Operative hysteroscopy will be performed at room temperature distention medium.
  Interventions: Procedure: Operative Hysteroscopy 24 Centigrade Degree
- 37 Centigrade Degree (Active Comparator): Operative hysteroscopy will be performed using a heated distention medium.
  Interventions: Procedure: Operative Hysteroscopy 37 Centigrade Degree

INTERVENTIONS:
Procedure: Operative Hysteroscopy 24 Centigrade Degree — Operative hysteroscopy will be performed at room temperature distention medium.
  Arms: 24 Centigrade Degree
Procedure: Operative Hysteroscopy 37 Centigrade Degree — Operative hysteroscopy will be performed using a heated distention medium.
  Arms: 37 Centigrade Degree

SUMMARY:
Minimally invasive applications are seen as the gold standard in today's gynecology practice and are frequently preferred by both patients and physicians. Less pain, shorter hospital stays, and better cosmetic results brought about by minimally invasive applications further increase their preference. One of these approaches is hysteroscopic interventions. Although hysteroscopy is a well-defined method, current research has focused on further reduction of pain. One of these methods is to warm the distention media at body temperature. theTaim of this study was to examine the effect of distention medium temperature on image quality, hyponatremia risk, and post-operative pain in operative hysteroscopy.

DETAILED DESCRIPTION:
Minimally invasive applications are seen as the gold standard in today's gynecology practice and are frequently preferred by both patients and physicians. Less pain, shorter hospital stays, and better cosmetic results brought about by minimally invasive applications further increase their preference. One of these approaches is hysteroscopic interventions. Although hysteroscopy is a well-defined method, current research has focused on further reduction of pain. One of these methods is to warm the distention media at body temperature.

The optimum distention medium temperature has not been determined in the "Best Practice in Outpatient Hysteroscopy Green Top Guideline" organized by The Royal College of Obstetricians and Gynecologists and "Guideline on Management of Fluid Distension Media in Operative Hysteroscopy" organized by the European Society of Gynecological Endoscopy. In routine practice, some physicians use distention fluid at room temperature, while others use it by warming it at body temperature. It is known that colder fluids cause irregular contractions in the uterus. In prospective studies, the effects of heating distention media at body temperature on pain were reported inconsistently. As clear data could not be obtained, the risk of further intravasation and hyponatremia that may occur with the image quality and, more importantly, the heating of the fluid was ignored. But; Freitas Fonseca et al. In his in vitro study in Brazil, it was shown by theoretical calculations that heating hysteroscopy irrigation fluids from 270C to 370C increased intravasation by 53%.

In light of the literature, and based on the ideas and possible risks in question, the aim of this study was to examine the effect of distention medium temperature on image quality, hyponatremia risk, and post-operative pain in operative hysteroscopy.

ELIGIBILITY:
Inclusion Criteria:

* To be planned for operative hysteroscopy due to an endometrial polyp or type 0-1 myoma in the range of 2-3 cm
* Having a vaginal delivery at least once before
* Ability to communicate adequately in Turkish or English

Exclusion Criteria:

* Pregnancy
* Active vaginal, and cervical infection

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Post-operative pain | 3 hours
  Post operative pain will evalute with numeric pain rating scale
  The scale is scored from 0 to 10. 0 means no pain and 10 means the most severe pain experienced.

SECONDARY OUTCOMES:
Post operavite Na Value Change | 1 minute
  Post-operative blood Na value will be checked.

CONTACTS AND LOCATIONS:
Overall Officials: Sabahattin A Ari, Asst. Prof., Principal Investigator — Izmir Bakircay University
Locations (1):
- Sabahattin Anil Ari, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
IPD will not be published.